CLINICAL TRIAL: NCT02937116
Title: An Open-Label, Multicenter Study of IBI308 in Subjects With Selected Advanced Solid Tumors
Brief Title: First in Human Study of IBI308 in Chinese Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308A101
Record Dates: First submitted 2016-10-08; First posted 2016-10-18 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Cancer, Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Phase 1a (Experimental): Participants will receive IBI308 1mg/kg, 3mg/kg or 10mg/kg intravenous every 2 weeks, or 200mg intravenous every 3 weeks and will be continued until disease progression or unacceptable toxicity.
  Drug: IBI308
  Interventions: Drug: IBI308
- Phase 1b Cohort A (Experimental): Participants will receive IBI308 200mg intravenous every 3 weeks and will be continued until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308
  Interventions: Drug: IBI308
- Phase 1b Cohort B (Experimental): Participants will receive IBI308 200mg intravenous every 3 weeks and will be continued until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308
  Interventions: Drug: IBI308
- Phase 1b Cohort C (Experimental): Participants will receive IBI308 200mg intravenous every 3 weeks and will be continued until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308
  Interventions: Drug: IBI308
- Phase 1b Cohort D (Experimental): Participants will receive IBI308 200mg in combination with cisplatin 75mg/m2 and pemetrexed 500mg/m2 intravenously every 3 weeks for upto 4 cycles, and those who haven't progressed will receive maintenance treatment of IBI308 200mg in combination with pemetrexed 500mg/m2 intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308/Cisplatinum/Pemetrexed
  Interventions: Drug: IBI308\Cisplatinum\Pemetrexed
- Phase 1b Cohort E (Experimental): Participants will receive IBI308 200mg and cisplatin 75mg/m2 intravenously every 3 weeks in combination with gemcitabine 1250mg/m2 intravenously day 1 and 8 of every 3 weeks for upto 6 cycles, and those those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308\gemcitabine\cisplatin
  Interventions: Drug: IBI308\cisplatin\gemcitabine
- Phase 1b Cohort F (Experimental): Participants will receive IBI308 200mg and oxaliplatin 130mg/m2 intravenously every 3 weeks in combination with capecitabine 1000mg/m2 orally day 1 to 14 of every 3 weeks for upto 6 cycles, and those those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308\oxaliplatin\capecitabine
  Interventions: Drug: IBI308\oxaliplatin\capecitabine
- Phase 1b Cohort G (Experimental): Participants will receive IBI308 200mg in combination with cisplatin 75mg/m2 intravenously and etoposide 100mg/m2 intravenously day 1 to 3 of every 3 weeks for upto 6 cycles. Those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308\etoposide\cisplatin
  Interventions: Drug: IBI308\etoposide\cisplatin
- Phase 1b Cohort H (Experimental): Participants will receive IBI308 200mg in combination with irinotecan 125mg/m2 intravenously day 1and 8 and 5-FU 1000mg/m2 intravenously day 1 to 3 of every 3 weeks for upto 6 cycles.Those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
  Drug: IBI308\irinotecan\5-FU
  Interventions: Drug: IBI308\irinotecan\5-FU

INTERVENTIONS:
Drug: IBI308
  Arms: Phase 1a; Phase 1b Cohort A; Phase 1b Cohort B; Phase 1b Cohort C
Drug: IBI308\Cisplatinum\Pemetrexed
  Arms: Phase 1b Cohort D
Drug: IBI308\cisplatin\gemcitabine
  Arms: Phase 1b Cohort E
Drug: IBI308\oxaliplatin\capecitabine
  Arms: Phase 1b Cohort F
Drug: IBI308\etoposide\cisplatin
  Arms: Phase 1b Cohort G
Drug: IBI308\irinotecan\5-FU
  Arms: Phase 1b Cohort H

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of IBI308 monotherapy or in combination with chemotherapy in patients with certain types of advanced solid tumors. Another purpose is to determine the pharmacokinetics, pharmacodynamics and immunogenicity of IBI308.

DETAILED DESCRIPTION:
This is a study which consists of phase 1a study (dose escalation stage) and phase 1b study (expansion stage). Phase 1a study will adopt the classical 3+3 dose escalation design, exploring safety and tolerance of 4 dose cohorts (1mg/kg, 3mg/kg, 200mg and 10mg/kg) and determining the recommended dose for phase 1b study. Phase 1b is expansion study of 8 cohorts which will evaluate anti-tumor efficacy and safety of eight IBI308 monotherapy or in combination with chemotherapy. Cohort A is IBI308 monotherapy for advanced melanoma. Cohort B is IBI308 monotherapy for advanced digestive system carcinoma or neuroendocrine neoplasm after failure or intolerance of first line standard therapy. Cohort C is IBI308 monotherapy for advanced non-small cell lung cancer (NSCLC) after failure or intolerance of first line standard therapy. Cohort D is IBI308 in combination with cisplatin and pemetrexed for treatment naïve locally advanced, recurrent or metastatic non-squamous NSCLC. Cohort E is IBI308 in combination with gemcitabine and cisplatin for treatment-naïve locally advanced, recurrent or metastatic squamous NSCLC. Cohort F is IBI308 in combination with oxaliplatin and capecitabine for treatment naïve locally advanced gastric or gastroesophageal junction adenocarcinoma. Cohort G is IBI308 in combination with etoposide and cisplatin for treatment naïve locally advanced, recurrent or metastatic high grade(G3) neuroendocrine tumor. Cohort H is IBI308 in combination with irinotecan and 5-FU for advanced high grade(G3) neuroendocrine tumor after failure of first line standard therapy. Phase 1a and 1b consist of screening period (28 days before enrollment), treatment period and follow up period (every 3 months until death or the end of study). In phase 1a, dose limiting toxicity (DLT) will be recorded for up to 28 days after the 1st dose of IBI308. Efficacy will be evaluated by RECIST v1.1. Adverse events will be monitored throughout the study. Further exploration of pharmacokinetic/pharmacodynamics and immunogenicity information will be assessed throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status grade 0 or 1
* Adequate bone marrow, liver, and renal function defined as: 1) Absolute neutrophil count >= 1.5* 10^9 cells/litre (L); 2) Platelets >=100 x 10^9 cells/L; 3) Hemoglobin >= 9 gram/deciliter (g/dL); 4) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 * upper limit of normal (ULN) for participants without hepatic cell cancer and hepatic metastasis, ALT and AST <= 5 * ULN for participants with hepatic cell cancer or hepatic metastasis; 5) Total bilirubin (TBIL) < 1.5 * ULN for participants without hepatic cell cancer, hepatic metastasis and confirmed/suspicious Gilbert syndrome, TBIL < 3 * ULN for participants with hepatic cell cancer, hepatic metastasis or confirmed/suspicious Gilbert syndrome; 6) Creatinine determined by serum creatinine levels <=1.5 * ULN or a calculated creatinine clearance of >= 50 mL/min/1.73 m^2; 7) urine protein -~+, 24 hour urine < 1 gram for participants with urine protein ++ or above; 8) activated partial thromboplastin time and international normalized ratio <= 1.5 * ULN; 9) thyroid stimulating hormone and free thyroxine 4 within normal range
* Tumor type

  * Phase 1a: advanced solid tumors after failure of standard therapy
  * Phase 1b Cohort A: cytologically or histologically confirmed advanced melanoma
  * Phase 1b Cohort B: cytologically or histologically confirmed advanced malignancies of the digestive system after failure of at least 1 line of standard therapy
  * Phase 1b Cohort C: cytologically or histologically confirmed advanced NSCLC without known epithelial growth factor receptor (EGFR) mutation and anaplastic lymphoma kinase (ALK) rearrangement after failure of 1st line standard therapy
  * Phase 1b Cohort D: treatment naive cytologically or histologically confirmed inoperable locally advanced (stage IIIB) or advanced (stage IV) nsNSCLC without known EGFR mutation and ALK rearrangement, participants with disease recurrence or progression within 6 months after completion of prior platinum doublet-based chemotherapy regimen as neoadjuvant or adjuvant therapy are not eligible
  * Phase 1b Cohort E: Cytologically or histologically confirmed, treatment naïve locally advanced, recurrent or metastatic squamous NSCLC without known EGFR mutation and ALK rearrangement. Participants with Stage IIIB NSCLC who progressed within 6 months after completion of platinum-based chemotherapy are not eligible.
  * Phase 1b Cohort F: Histologically confirmed locally advanced, recurrent or metastatic gastric or esophagogastric junction adenocarcinoma without known HER2 amplification.
  * Phase 1b Cohort G: Cytologically or histologically confirmed, treatment naïve locally advanced, recurrent or metastatic high grade(G3) neuroendocrine tumor with Ki-67>20%.
  * Phase 1b Cohort H: Cytologically or histologically confirmed advanced high grade(G3) neuroendocrine tumor with Ki-67>20% after failure of first line standard therapy. Participants progressed within 6 months after completion of adjuvant or neoadjuvant chemotherapy are eligible.
* At least 1 measurable site of disease per RECIST v1.1

Exclusion Criteria:

* Prior treatment of any antibody of PD-1 or PD-L1
* Prior treatment of ipilimumab, unless all the following requirements are met:

  * Full resolution of ipilimumab related adverse effects (including immune related adverse effects) and no treatment for these adverse events (AEs) for at least 4 weeks prior to the time of enrollment
  * Minimum of 12 weeks from the first dose of ipilimumab and >6 weeks from the last dose
  * No history of severe immune related adverse effects from ipilimumab (CTCAE Grade 4; CTCAE Grade 3 requiring treatment >4 weeks)
  * Unequivocal PD following a dose of ipilimumab
* HIV infection
* Active HBV or HCV infection
* Uncontrolled complication including but not limited to :

  * Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias or congestive heart failure
  * History of stroke, myocardial infarction or intracranial hemorrhage within 6 months prior to the enrolment
* History or risk of autoimmune disease
* Known interstitial lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The fifth medical center of the PLA general hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jiang H, Zheng Y, Qian J, Mao C, Xu X, Li N, Xiao C, Wang H, Teng L, Zhou H, Wang S, Zhu D, Peng B, Shen L, Xu N. Safety and efficacy of sintilimab combined with oxaliplatin/capecitabine as first-line treatment in patients with locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma in a phase Ib clinical trial. BMC Cancer. 2020 Aug 14;20(1):760. doi: 10.1186/s12885-020-07251-z. PMID 32795349
- [Result] Jiang H, Zheng Y, Qian J, Mao C, Xu X, Li N, Xiao C, Wang H, Teng L, Zhou H, Wang S, Zhu D, Sun T, Yu Y, Guo W, Xu N. Efficacy and safety of sintilimab in combination with chemotherapy in previously untreated advanced or metastatic nonsquamous or squamous NSCLC: two cohorts of an open-label, phase 1b study. Cancer Immunol Immunother. 2021 Mar;70(3):857-868. doi: 10.1007/s00262-020-02738-x. Epub 2020 Oct 17. PMID 33070260
- [Derived] Wei J, Lu X, Liu Q, Fu Y, Liu S, Li L, Liu F, Fan X, Yang J, Yang Y, Zhao Y, Guan W, Liu B. Efficacy and Safety of Sintilimab in Combination with Concurrent Chemoradiotherapy for Locally Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (SHARED): Study Protocol of a Prospective, Multi-Center, Single-Arm Phase 2 Trial. Cancer Manag Res. 2022 Jun 17;14:2007-2015. doi: 10.2147/CMAR.S355687. eCollection 2022. PMID 35747712
- [Derived] Jia R, Li Y, Xu N, Jiang HP, Zhao CH, Liu RR, Shi Y, Zhang YY, Wang SY, Zhou H, Xu JM. Sintilimab in Patients with Previously Treated Metastatic Neuroendocrine Neoplasms. Oncologist. 2022 Aug 5;27(8):e625-e632. doi: 10.1093/oncolo/oyac097. PMID 35647908
- [Derived] Jiang H, Li N, Wang H, Chen Z, Zheng Y, Qian J, Mao C, Xu X, Xiao C, Zhang X, Zhou H, Wang S, Chen W, Yin X, Sun J, Peng B, Teng L, Xu N. Assessment of TMB, PD-L1, and lymphocyte to monocyte ratio as predictive potential in a phase Ib study of sintilimab in patients with advanced solid tumors. Am J Cancer Res. 2021 Sep 15;11(9):4259-4276. eCollection 2021. PMID 34659886
- [Derived] Zhang J, Wu L, Liu J, Lin M. A metastatic intrahepatic cholangiocarcinoma treated with programmed cell death 1 inhibitor: a case report and literature review. Immunotherapy. 2020 Jun;12(8):555-561. doi: 10.2217/imt-2019-0100. Epub 2020 May 6. PMID 32372672
- See also: Abstract for Cohort E on Jtho.2018 — https://doi.org/10.1016/j.jtho.2018.10.018

RESULTS

PARTICIPANT FLOW:
Groups:
- Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1): 1mg/kg intravenous Q2W, will be continued until disease progression or unacceptable toxicity.
- Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2): 3mg/kg intravenous Q2W, will be continued until disease progression or unacceptable toxicity.
- Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3): 10mg/kg intravenous Q2W, will be continued until disease progression or unacceptable toxicity.
- Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4): 200mg intravenous Q3W, will be continued until disease progression or unacceptable toxicity.
- MEL: Sintilimab 200mg Q3W (Cohort A); Malignant Tumor of the Digestive System or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B); NSCLC: Sintilimab 200mg Q3W (Cohort C): Subjects received sintilimab 200mg intravenous every 3 weeks and will be continued until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
- nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D): Subjects received sintilimab 200mg in combination with cisplatin 75mg/m2 and pemetrexed 500mg/m2 intravenously every 3 weeks for upto 4 cycles, and those who haven't progressed will receive maintenance treatment of IBI308 200mg in combination with pemetrexed 500mg/m2 intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
- scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E): Subjects received sintilimab 200mg and cisplatin 75mg/m2 intravenously every 3 weeks in combination with gemcitabine 1250mg/m2 intravenously day 1 and 8 of every 3 weeks for upto 6 cycles, and those those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
- Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F): Subjects received sintilimab 200mg and oxaliplatin 130mg/m2 intravenously every 3 weeks in combination with capecitabine 1000mg/m2 orally day 1 to 14 of every 3 weeks for upto 6 cycles, and those those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
- Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G): Subjects received sintilimab 200mg in combination with Cisplatin 75mg/m2 intravenously Day 1 and Etoposide 100mg/m2 intravenously Day 1-3 every 3 weeks for upto 6 cycles, and those those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
- Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H): Subjects received sintilimab 200mg intravenously Day 1 in combination with Irinotecan 125mg/m2 intravenously Day 1 and 8, and 5-FU 1000mg/m2 intravenously Day 1-3 every 3 weeks for upto 6 cycles, and those those who haven't progressed will receive maintenance treatment of IBI308 200mg intravenously every 3 weeks until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
Period: Overall Study
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor of the Digestive System or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Started | 3 | 3 | 3 | 3 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor of the Digestive System or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7 | 233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.33 (17.010) | 46 (15.524) | 48 (6.557) | 50 (16.093) | 49.13 (13.061) | 52.27 (11.280) | 55.35 (11.201) | 60.52 (6.539) | 62.30 (6.951) | 58.20 (8.600) | 62.86 (4.140) | 49.29 (11.912) | 54.54 (11.291)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 1 | 7 | 30 | 6 | 5 | 1 | 2 | 1 | 2 | 61
  Male | 2 | 1 | 0 | 2 | 15 | 57 | 31 | 16 | 19 | 18 | 6 | 5 | 172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 3 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7 | 233
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 3 | 3 | 3 | 3 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7 | 233

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-limiting Toxicities (DLTs)
Time Frame: Up to 28 days in Cycle 1
Population: All participants in Parts A1 to A4 who received ≥1 dose of study treatment and either 1) had a DLT in Cycle 1 or 2) received ≥90% of the prescribed dose of Sintilimab in Cycle 1 and completed all safety evaluations ≥28 days after the first administration of Sintilimab without experiencing DLT. Per protocol, cohort A to H were not analyzed.
Measure: Number; unit: Participants
Groups:
- Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B); NSCLC: Sintilimab 200mg Q3W (Cohort C): Subjects received sintilimab 200mg intravenous every 3 weeks and will be continued until disease progression or unacceptable toxicity or withdrawal of informed consent or up to 24 months of treatment.
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |

2. Primary Outcome: Number of All Study Participants Who Demonstrate a Tumor Response
Time Frame: Through out the study (up to 2 years)
Measure: Number; unit: Participants
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
Participants | 0 | 1 | 0 | 1 | 1 | 13 | 5 | 13 | 11 | 17 | 3 | 1

3. Primary Outcome: Objective Response Rate (ORR) According to RECIST 1.1 as Assessed by Independent Review Committee by Investigator
Description: ORR was defined as the percentage of participants in the analysis population who had achieved BOR of CR or PR according to RECIST 1.1.
Time Frame: Through out the study (up to 2 years)
Population: Participants from cohort A to H that received ≥1 dose of study treatment. Per protocol, Part A1 to A4 (dose-escalation) was not analyzed for efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
percentage of participants |  |  |  |  | 4.5 [0.1 to 22.8] | 14.9 [8.2 to 24.2] | 13.5 [4.5 to 28.8] | 61.9 [38.4 to 81.9] | 55.0 [31.5 to 76.9] | 85.0 [62.1 to 96.8] | 42.9 [9.9 to 81.6] | 14.3 [0.4 to 57.9]

4. Secondary Outcome: PFS According to RECIST 1.1 as Assessed by Investigator
Time Frame: Through out the study (up to 2 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
Days |  |  |  |  | 62.0 [59.0 to 125.0] | 66.0 [64.0 to 95.0] | 84.0 [60.0 to 187.0] | 377.0 [92.0 to NA] — PFS range upper limit of 95% CI not reached | 194.0 [160.0 to 239.0] | 230.0 [189.0 to 287.0] | NA [NA to NA] — Median PFS and PFS range lower and upper limit of 95% CI not reached (no disease progression by last progression assessment) | NA [68.0 to NA] — Median PFS and PFS range upper limit of 95% CI not reached

5. Secondary Outcome: DOR According to RECIST 1.1 as Assessed by Investigator
Time Frame: Through out the study (up to 2 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
Days |  |  |  |  | NA [NA to NA] — Median DOR and DOR lower and upper limit not reached | NA [86.0 to NA] — Median DOR and DOR upper limit not reached (no progressive disease by time of last disease assessment) | 368.0 [190.0 to NA] — DOR upper limit not reached | NA [NA to NA] — Median DOR and DOR lower and upper limit not reached | 170.5 [58.0 to NA] — DOR upper limit not reached | 181.0 [146.0 to 221.0] | NA [NA to NA] — Median DOR and DOR lower and upper limit of 95% CI not reached | NA [NA to NA] — Median DOR and DOR lower and upper limit of 95% CI not reached

6. Secondary Outcome: TTR According to RECIST 1.1 as Assessed by Investigator
Time Frame: Through out the study (up to 2 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
Days |  |  |  |  | 63.0 [NA to NA] — TTR louwer and upper limit not reached | 64.0 [61.0 to 70.0] | 63.0 [60.0 to 189.0] | 63.0 [62.0 to 120.0] | 62.0 [58.0 to 68.0] | 63.0 [62.0 to 65.0] | 62.0 [62.0 to 63.0] | 62.0 [62.0 to 62.0]

7. Secondary Outcome: OS for Participants
Time Frame: Through out the study
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 87 | 37 | 21 | 20 | 20 | 7 | 7
Days |  |  |  |  | 518.0 [349.0 to NA] — OS range upper limit not reached | 342.0 [218.0 to 441.0] | 431.0 [196.0 to 562.0] | 566.0 [158.0 to NA] — OS range upper limit not reached | 461.0 [308.0 to NA] — OS range upper limit not reached | NA [287.0 to NA] — Median OS and OS range upper limit not reached | NA [NA to NA] — Median OS and OS range lower and upper limit of 95% CI not reached (no death by last assessment) | NA [NA to NA] — Median OS and OS range lower and upper limit of 95% CI not reached (no death by last assessment)

8. Secondary Outcome: Area Under the Concentration-time Curve From Zero Time (Predose) to the Time of the Last Measurable Concentration (AUC0-t)
Time Frame: Cycle 1: pre-dose, post-dose at 0, 1, and 6 hours, and Days 2, 3, 8, 15, and 22, and 29
Population: All participants in Parts A1 to A4 receiving a single dose of drug during Cycle 1 (28 days) and having available AUC 0-t data. Per protocol, participants in cohort A to H were not included in the escalating dose PK analysis..
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/ml
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
h*ug/ml | 4800 (8.2) | 12300 (35.2) | 39800 (14.5) | 10800 (49.3) |  |  |  |  |  |  |  |

9. Secondary Outcome: Maximum Concentration (Cmax) of Sintilimab in Solid Tumor Participants
Time Frame: Cycle 1: pre-dose, post-dose at 0, 1, 6 hours, and Days 2, 3, 8, 15, and 22, and 29
Population: All participants in Parts A1 to A4 receiving a single dose of drug during Cycle 1 (28 days) and having available Cmax data. Per protocol, participants in cohort A to H were not included in the escalating dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ug/ml | 21.9 (11.3) | 69.7 (12.2) | 220 (13.4) | 54.6 (50.5) |  |  |  |  |  |  |  |

10. Secondary Outcome: Time to Maximum Concentration (Tmax) of Sintilimab in Solid Tumor Participants
Time Frame: Cycle 1: pre-dose, post-dose at 0, 1, 6 hours, and Days 2, 3, 8, 15, and 22, and 29
Population: All participants in Parts A1 to A4 receiving a single dose of drug during Cycle 1 (28 days) and having available Tmax data. Per protocol, participants in cohort A to H were not included in the escalating dose PK analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hours | 1.05 [1.05 to 1.08] | 2.07 [2.07 to 2.08] | 2.27 [1.10 to 2.33] | 1.93 [1.08 to 2.13] |  |  |  |  |  |  |  |

11. Secondary Outcome: The Half-life (t1/2) of IBI308 in Plasma After Single Dose Administration
Time Frame: Cycle 1: pre-dose, post-dose at 0, 1, 6 hours, and Days 2, 3, 8, 15, and 22, and 29
Population: All participants in Parts A1 to A4 receiving a single dose of drug during Cycle 1 (28 days) and having available T1/2 data. Per protocol, participants in cohort A to H were not included in the escalating dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Days | 17 (7.3) | 12.7 (44.6) | 12.5 (26.4) | 16.1 (32.6) |  |  |  |  |  |  |  |

12. Secondary Outcome: Volume of Distribution of IBI308 in Plasma After Single Dose Administration
Time Frame: Cycle 1: pre-dose, post-dose at 0, 1, 6 hours, and Days 2, 3, 8, 15, and 22, and 29
Population: All participants in Parts A1 to A4 receiving a single dose of drug during Cycle 1 (28 days) and having available volume of distribution data. Per protocol, participants in cohort A to H were not included in the escalating dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
L | 5.02 (24.0) | 5.14 (18.7) | 5.95 (10.5) | 7.2 (45.0) |  |  |  |  |  |  |  |

13. Secondary Outcome: Clearance of IBI308 in Plasma After Single Dose Administration
Time Frame: Cycle 1: pre-dose, post-dose at 0, 1, 6 hours, and Days 2, 3, 8, 15, and 22, and 29
Population: All participants in Parts A1 to A4 receiving a single dose of drug during Cycle 1 (28 days) and having available clearance data. Per protocol, participants in cohort A to H were not included in the escalating dose PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml/h
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ml/h | 8.53 (20.7) | 11.7 (33.3) | 13.7 (15.9) | 12.9 (61.1) |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Up to approximately 90 days (through Final Database cut-off date of 30-Oct-2017) for Phase Ia (Part A1 to A4); Up to approximately 90 days (through Final Database cut-off date of 17-Apr-2019) for Phase Ib (Cohort A to F); Up to approximately 90 days (through Final Database cut-off date of 30-Sep-2019) for Phase Ib (Cohort G to H);
Description: All adverse events, including serious adverse events, will be collected since the consent form is signed until 90th day after last administration of investigation products, either observed by investigator or by the spontaneous reported by subjects.
Arm/Group | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) | MEL: Sintilimab 200mg Q3W (Cohort A) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) | NSCLC: Sintilimab 200mg Q3W (Cohort C) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H)
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/3 | 3/3 | 1/3 | 12/22 | 57/87 | 25/37 | 9/21 | 8/20 | 3/20 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/3 | 1/3 | 0/22 | 18/87 | 11/37 | 3/21 | 9/20 | 6/20 | 2/7 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 18/22 | 82/87 | 35/37 | 19/21 | 20/20 | 20/20 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) (N=3) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) (N=3) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) (N=3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) (N=3) | MEL: Sintilimab 200mg Q3W (Cohort A) (N=22) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) (N=87) | NSCLC: Sintilimab 200mg Q3W (Cohort C) (N=37) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) (N=21) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) (N=20) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) (N=20) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) (N=7) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H) (N=7)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyopneumothorax (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal hydrocele (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Solid Tumors: Sintilimab 1mg/kg Q2W (Part A1) (N=3) | Solid Tumors: Sintilimab 3mg/kg Q2W (Part A2) (N=3) | Solid Tumors: Sintilimab 10mg/kg Q2W (Part A3) (N=3) | Solid Tumors: Sintilimab 200mg/kg Q3W (Part A4) (N=3) | MEL: Sintilimab 200mg Q3W (Cohort A) (N=22) | Malignant Tumor or Neuroendocrine Tumor: Sintilimab 200mg Q3W (Cohort B) (N=87) | NSCLC: Sintilimab 200mg Q3W (Cohort C) (N=37) | nsNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort D) (N=21) | scNSCLC: Sintilimab 200mg Q3W + Chemotherapy (Cohort E) (N=20) | Gastric or Gastroesophageal Junction Adenocarcinoma: Sintilimab 200mg Q3W + Chemotherapy (Cohort F) (N=20) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort G) (N=7) | Neuroendocrine Tumors: Sintilimab 200mg Q3W + Chemotherapy (Cohort H) (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 2 | 37 | 10 | 9 | 17 | 12 | 6 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 8 | 1 | 1 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 0 | 1 | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 2 | 4 | 2 | 1 | 2 | 6 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 6 | 1 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 2 | 10 | 4 | 3 | 2 | 2 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 4 | 2 | 2 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9 | 8 | 3 | 2 | 6
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 7 | 6 | 3 | 2 | 4
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 1 | 23 | 5 | 7 | 5 | 2 | 1 | 4
Chest discomfort (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 2 | 1 | 4 | 15 | 6 | 6 | 6 | 3 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 7 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sebaceous gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 0 | 1 | 0 | 5 | 3 | 2 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 3 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 1 | 3 | 22 | 7 | 7 | 1 | 5 | 0 | 3
Amylase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 3 | 5 | 28 | 6 | 6 | 2 | 5 | 2 | 4
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 2 | 3 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 1 | 5 | 14 | 2 | 0 | 1 | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 1 | 1 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 4 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 5 | 3 | 6 | 2 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 2 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 2 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram low voltage (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 8 | 10 | 4 | 4 | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Granulocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 10 | 3 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0 | 2 | 5 | 3 | 10 | 16 | 10 | 5 | 4
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 7 | 2 | 2 | 14 | 16 | 2 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Procalcitonin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Thyroid function test abnormal (Investigations) | 2 | 1 | 0 | 1 | 0 | 18 | 0 | 0 | 1 | 3 | 1 | 1
Thyroxine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thyroxine free decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thyroxine free increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Thyroxine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Tri-iodothyronine decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Tri-iodothyronine free increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 6 | 5 | 1 | 3 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 5 | 14 | 4 | 7 | 18 | 10 | 5 | 5
White blood cell count increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 5 | 6 | 8 | 8 | 2 | 3 | 6
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 5 | 3 | 2 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 7 | 2 | 0 | 0 | 0 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 14 | 5 | 1 | 5 | 0 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 10 | 1 | 1 | 0 | 0 | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 11 | 2 | 1 | 2 | 3 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 10 | 4 | 1 | 2 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0 | 13 | 1 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 9 | 5 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 3 | 3 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 2 | 1 | 1 | 1 | 22 | 5 | 1 | 4 | 2 | 2 | 3
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 7 | 5 | 1 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 7 | 5 | 5 | 4 | 5 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 2 | 0 | 6 | 0 | 2 | 6 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT02937116/Prot_SAP_000.pdf